CLINICAL TRIAL: NCT06902038
Title: Clinical Research on the Use of Immune Checkpoint Inhibitors Combined With Chidamide for the Functional Cure of AIDS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jun Chen, MD (Other Government)
Responsible Party: Sponsor-Investigator, Jun Chen, MD, Deputy Director of Infection and Immunization, Shanghai Public Health Clinical Center
Organization: Shanghai Public Health Clinical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PD-1 inhibitor
Record Dates: First submitted 2025-02-25; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-02

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — Immune Checkpoint Inhibitors; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): Saline 50ml q3w ×2
  Interventions: Drug: Saline (NaCl 0,9 %) (placebo)
- Experimental sindilizumab (Experimental): 100mg of sindilizumab, was dissolved in 50ml normal saline, q3w was administered ×2
  Interventions: Drug: PD-1 inhibitor
- Experimental sindilizumab and sidarbenamide (Experimental): 100mg of sindilizumab, was dissolved into 50ml of normal saline q3w ×2+ sidarbenamide 10mg biw orally for 2 weeks
  Interventions: Drug: PD-1 inhibitor; Drug: Sidarbenamide

INTERVENTIONS:
Drug: PD-1 inhibitor — 100mg of sindilizumab, was dissolved into 50ml of normal saline q3w ×2
  Arms: Experimental sindilizumab; Experimental sindilizumab and sidarbenamide
Drug: Sidarbenamide — Sidarbenamide 10mg biw orally for 2 weeks
  Arms: Experimental sindilizumab and sidarbenamide
Drug: Saline (NaCl 0,9 %) (placebo) — Saline 50ml Q3W ×2
  Other Names: Placebo Comparator
  Arms: Control group

SUMMARY:
Evaluate the efficacy and safety of immune checkpoint inhibitors combined with chidamide as an "activate and kill" strategy to extend viral rebound time, reduce the HIV reservoir, and achieve functional cure.

DETAILED DESCRIPTION:
This project plans to conduct a prospective randomized controlled study, using immune checkpoint inhibitors combined with chidamide, while applying antiretroviral therapy interruption(ATI) to further enhance the immune killing effect of this strategy, with the aim of accelerating the clearance of the HIV reservoir and delaying the time of viral rebound, thereby achieving a functional cure for AIDS.

ELIGIBILITY:
Inclusion Criteria:

* People diagnosed with HIV infection;
* Age ≥18 years old;
* General good health, body mass index ≥18.0 to <35.0 kg/m2;
* Able and willing to comply with the time requirements for research visits and evaluations;
* have received ART therapy for at least 24 months, and plasma HIV-1 RNA < 50 copies /ml for two consecutive times with a time interval of at least 12 months;
* During the screening period, the number of CD4+ T cells was ≥350 cells /μl(including boundary values);
* Agree to adhere to contraception during the course of participating in the project and within 6 months after the end of the trial;
* Willing to sign informed consent

Exclusion Criteria:

* Have suffered from any serious acute disease within 8 weeks;
* Subjects with a history of active autoimmune disease or autoimmune disease requiring systemic treatment;
* Pre-treatment/exposure to any other immune checkpoint inhibitor [e.g., anti-programmed cell death protein 1(PD-1), anti-PD-L1, anti-PD-L2, anti-CTLA4, etc.].
* The patient has received the following treatment:

  1. Received other anti-latency drugs within 30 days prior to enrollment;
  2. Radiotherapy or chemotherapy 30 days before screening;
  3. Immunosuppressive therapy 60 days before screening;
  4. Treatment with immunomodulators (e.g., interleukin, interferon), hydroxyurea, or phosphonic acid 60 days prior to screening
  5. Receiving HIV vaccine or systemic cytotoxic chemotherapy 60 days before screening;
  6. Previous immunoglobulin (IgG) therapy
  7. Received blood transfusion or cell growth factor therapy in the 90 days prior to screening
  8. Drugs such as rifampicin and rifambutin were being used at the time of screening or at the planned treatment stage;
* Laboratory tests meet the following standards:

  1. Absolute neutrophil count (ANC) < 1.50×109/L; Hemoglobin (Hb) < 105g/L(male) or < 95g/L(female); Platelet < 75×109/μL; International Normalized Ratio (INR) > 1× Upper Limit of Normal (ULN)
  2. Serum alanine aminotransferase (ALT) > 1.5× upper limit of normal (ULN), serum aspartate aminotransferase (SGOT/AST) > 1.5× upper limit of normal (ULN), total bilirubin, direct bilirubin > 1.5× upper limit of normal (ULN), serum creatinine > 1.5× upper limit of normal (ULN), And the abnormality has clinical significance;
  3. Five abnormalities of thyroid function with clinical significance: test items include triiodothyronine (T3), tetraiodothyronine (T4), free triiodothyronine (FT3), free tetraiodothyronine (FT4), and thyroid stimulating hormone (TSH).
  4. The epinephrine test was abnormal and clinically significant;
  5. Blood glucose and glycated hemoglobin were abnormal and clinically significant
* Twelve-lead electrocardiogram was abnormal and clinically significant at the time of enrollment;
* Interstitial changes were detected by chest CT at the time of enrollment;
* Subjects with severe heart disease, symptomatic or asymptomatic arrhythmia;
* Patients with co-infection such as HBV, HCV, syphilis, diabetes, and other liver diseases;
* Subjects with a history of active or suspected malignancy or malignancy (other than basal cell skin cancer or cervical cancer in situ) within five years.
* Subjects with a history of tuberculosis or active tuberculosis.
* Subjects with psychiatric or substance abuse disorders known to interfere with the requirements of the experiment.
* Subjects who received immunomodulatory or immunosuppressive therapy in the 24 weeks prior to first taking the study drug.
* Pregnant and lactating women;
* Mental illness or drug abuse interferes with the conduct of the test.
* Histone deacetylase inhibitors, such as valproic acid, butyrate, phenyl butyrate, etc., but can be included after a 28-day washout period;
* Patients with severe cardiac insufficiency [New York College of Cardiology (NYHA) Grade IV for cardiac insufficiency];
* any arterial thromboembolism event, including myocardial infarction, unstable angina pectoris, cerebrovascular accident, or transient ischemic attack, occurred within 6 months prior to treatment induction; Standardized treatment of uncontrolled hypertension (systolic blood pressure ≥150mmHg or diastolic blood pressure ≥100mmHg); Cardiomyopathy;
* Patients had significant QT/QTC intervals during the screening period (Fridericia formula: QTcF=QT/RR0.33) prolonged (e.g., repeated measurements show a QTc interval >450 ms, or there is another risk of torsive ventricular TdP [e.g., heart failure, hypokalemia, familial long QT syndrome]) or combined use of drugs that may cause a prolonged QT/QTc interval;
* Allergic or anti-drug antibodies to the drug or excipient used in this test are known.

The researchers judged that they were not suitable to participate in this experiment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-03-22 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Time interval from antiretroviral therapy interruption to antiretroviral treatment restart | From baseline to the date of antiretroviral treatment restart, up to 12 weeks

SECONDARY OUTCOMES:
The ratio of HIV RNA<50 copies /ml was maintained at 12 weeks | 12 weeks
Changes in HIV DNA levels from baseline to antiretroviral treatment restart | From baseline to the date of antiretroviral treatment restart, up to 12 weeks
Incidence of drug-related adverse events before antiretroviral treatment restart | From date of randomization to the date of antiretroviral treatment restart, up to 14 weeks.
Changes in HIV-specific CD8+ T response from baseline with Day8 and Day29 and ART restart | From baseline to Day 8, Day 29 and antiretroviral treatment restart, up to 12 weeks
Changes in PD-1 (+) CD4 T cells and CD8 T cells from baseline at Day8 and Day29 and ART restart | From baseline to Day 8, Day 29 and antiretroviral treatment restart, up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jun Chen, MD, Principal Investigator — Shanghai Public Health Clinical Center

IPD SHARING:
Plan to Share IPD: No